CLINICAL TRIAL: NCT01128010
Title: Role of CCL2 in Alcoholic Liver Diseases
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Other Study IDs: DD-CCL2
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2002-12

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- alcoholic liver disease: alcoholic liver disease patients undergoing a transjugular liver biopsy in our institution
- controls: Healthy controls patients recruited from the Occupational Medicine Department during a routine physical examination

SUMMARY:
Immune dysregulations, including cytokines and chemokines secretions occurs in alcoholic liver disease. Serum levels and liver expression of CCL2 are increased in patients with alcoholic hepatitis but the role of this chemokine in the pathogenesis of alcoholic liver disease is nevertheless unknown. The aim of the study is to analyze plasma level and liver expression of CCL2 and their relation with liver disease severity and inflammatory infiltrate in our cohort of alcoholic patients. We studied also the association between -2518 CCL2 polymorphism and the severity of alcoholic liver disease.

ELIGIBILITY:
ALD patients

Inclusion Criteria:

* Excess alcohol intake
* Abnormality of liver biopsy compatible with alcoholic aetiology
* Caucasian ethnicity

Exclusion Criteria:

* Presence of any other chronic liver disease
* co-infection with HIV Controls Inclusion criteria
* Caucasian ethnicity
* presence of a disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing transjugular liver biopsy for alcoholic liver disease will be include in the study to measure plasma levels and hepatic expression of CCL2. We determine also the rs1024611 polymorphism of these patients. All these parameters are correlated to severity of the disease.
  The frequency of the presence of this polymorphism was also compared to a population of healthy subjects.
Sampling Method: Probability Sample